CLINICAL TRIAL: NCT07369544
Title: The Effect of Preoperative Hugging With Family Members on Preoperative Anxiety Levels and Postoperative Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Balikesir Hospital Eduation and Research (Other Government)
Responsible Party: Principal Investigator, Sevgi Kutlusoy, ASSOCİATE PROF, University of Health Sciences Balikesir Hospital Eduation and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MTÜ-AAD-2025/154
Record Dates: First submitted 2025-12-31; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain Management; Anxiety; Non-Pharmacological Interventions
Keywords: Postoperative Pain Management; Anxiety; Non-Pharmacological Interventions
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hugging group (Active Comparator): Patients will be given the opportunity to hug family members for at least 20 seconds before the surgery.
  Interventions: Behavioral: Patients will be given the opportunity to hug family members for at least 20 seconds before the surgery.
- control group (Active Comparator): standard practice
  Interventions: Other: The standard anesthesia protocol will be followed

INTERVENTIONS:
Behavioral: Patients will be given the opportunity to hug family members for at least 20 seconds before the surgery. — Patients will be given the opportunity to hug family members for at least 20 seconds before the surgery.
  Arms: Hugging group
Other: The standard anesthesia protocol will be followed — The standard anesthesia protocol will be followed
  Arms: control group

SUMMARY:
The aim of this randomized prospective study is to examine the effect of preoperative family hugging (for at least 20 seconds) on preoperative anxiety levels and postoperative pain.

The main question the study aims to answer is:

* Does preoperative hugging reduce anxiety levels?
* Does preoperative hugging reduce postoperative pain scores? Anxiety and pain scores will be evaluated between patients who hugged and those who did not hug their family members before surgery, and whether hugging has an effect will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* ASA 1 and ASA-2 patients

Exclusion Criteria:

* emergency surgery
* malignancy surgery
* neurological and psychiatric illnesses
* chronic pain
* substance abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Does preoperative hugging reduce anxiety levels? | Preoperative STAI-I and STAI-II anxiety levels of patients will be measured. The relationship between the groups will be evaluated.
  Preoperative The State-Trait Anxiety Inventory (STAI) I and STAI-II anxiety levels of patients will be measured. This scale gives scores between 20 and 80. The significance of these differences between groups will be evaluated.
  A higher score indicates a higher anxiety level. The clinically significant score for STAI anxiety level is stated as 39-40.

SECONDARY OUTCOMES:
Does preoperative hugging reduce postoperative pain scores? | Postoperative NRS pain scores of patients at 30 minutes and 6 hours will be examined. The relationship between the groups will be evaluated.
  Postoperative NRS pain scores of patients at 30 minutes and 6 hours will be examined. It usually ranges from 0 to 10; 0 represents "no pain" and 10 represents "the most severe pain imaginable". The relationship between the groups will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Meah, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided